CLINICAL TRIAL: NCT06688474
Title: Otis Brux-Sensor Night Guard - a Novel Wireless Custom Night Guard System with Pressure Sensors to Quantitatively Measure Bite Compression Forces and Alleviate Sleep Bruxism
Brief Title: A Sensor-enhanced Mouth Guard to Quantitatively Measure Bite Compression Forces.
Status: Completed | Type: Observational
Sponsor: Otis Dental, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 1R43HL168988-01A1 (NIH)
Record Dates: First submitted 2024-11-08; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Bruxism, Sleep-Related
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bruxism Cohort: 2 male participants with diagnosed Bruxism will wear the device for 21 days, over a 6+ hour sleep period each night.

SUMMARY:
The goal of this study is to determine if the Otis Brux-Sensor Night Guard (OBSNG) can record the bite compression forces of participants with Bruxism. The main questions it aims to answer is:

1. Is it possible to design and miniaturize electrical hardware components small enough to fit onto the molar region of the custom night guard?
2. If successfully miniaturized, will we be able to capture bite compression force profiles and optimize data collection for analysis?

Participants would wear the device for 21 days, over a 6+ hour sleep period each night.

DETAILED DESCRIPTION:
Otis Dental proposes to develop the Otis Brux-Sensor Night Guard (OBSNG), which is a novel wireless custom night guard system with pressure sensors that can quantitatively measure bite compression forces during sleep (patent granted in June 2021). If successful, anyone suffering from Bruxism will have improved protection against the painful and damaging symptoms via a sensor-enhanced custom night guard. Dental providers can analyze and monitor bruxism compression force trends over time, thereby streamlining quality patient care through optimized treatment plans.

The technology is comprised of the Otis Custom Night Guard with an embedded electronics system that is coupled to a portion of the guard covering an axial plane of a tooth. The electronics system will be comprised of an antenna, capacitive sensor, microcontroller, and power supply. The sensor will produce and measure signals corresponding to bite compression forces generated by a wearer, over a period of time during sleep.

There are four key components to the innovation: (1) Otis Custom Night Guard. The Otis Custom Night Guard offers more comfort and protection from Bruxism compared to current products in the market (OTC and custom-made). After years of research and multiple rounds of pilot testing, Otis determined that their Custom Night Guard would be made with an equal ratio of hard co-polyester and soft polyurethane materials. In doing so, the soft inner liner would provide a level shock absorbance from jaw clenching, while the hard outer layer would provide protection against teeth grinding. It was also determined that making their custom night guards in a 2-3mm thickness, rather than the traditional 4-5mm thickness, would provide optimal comfort and user compliance. (2) Brux-Sensor. To generate the OBSNG, force-sensing resistors (FSRs) will be placed on either side of the posterior region of the Otis Custom Night Guard to collect optimal compression forces generated by jaw muscles around the Temporomandibular Joint. This sensor will allow for accurate measurements of the clenching forces applied by the patients over time. The force data can be measured at high frequencies in excess of once per second and stored in an onboard memory, allowing for a complete time-force profile for one night of usage. In the long term, an accelerometer will be integrated into the sensor to track sleep quality and jaw motion. Eventually, Otis will correlate this data to assess the patients' stress/anxiety level and establish relevant correlations with jaw forces and bruxism treatment plans. (3) Storage/Travel Case. Each OBSNG will come with a storage/travel case designed to store/protect the Otis custom night guard when not in use. The case will also act as a recharge station when not being used - enabling wireless charging and seamless data transferring to the Otis App for biofeedback. (4) Otis App. Otis will develop an app that allows patients to access personalized and regimented dental care tips and exercises that alleviate bruxism rates, dental wear and pain, headaches, shoulder tension, etc. (e.g., DIY jaw/head/ neck/shoulder massage videos). The app will also provide educational wellness information, instructional exercises to reduce stress levels and improve sleep quality (e.g., 4-7-8 breathing, meditation reminder, etc.), and discounts to partnering stress therapy apps (e.g., Noom, Headspace, Calm, etc.).

Participants will be recruited to test the OBSNG for 21 days, during 6+ hours of sleep. Upon completing the study and collecting all compression force data from each participant, the research team will begin averaging all compression force episodes throughout each of the 6+ hours of sleep per night and graph all 21 nights of averaged scores to show every participant's Bruxism pattern during the study. Upon successful build of a working prototype, the team will accomplish their first milestone by determining the bruxism severity (no/mild or mod/severe), based on the range of compression forces. The second milestone will be achieved by validating participants' bruxism severity through data points showing compression force.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years of age; male and/or female; healthy with exception to being diagnosed with Bruxism.

Exclusion Criteria:

* N/A

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: US participants only.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Analysis of Force Data for Bruxism Diagnosis | 21 Days
  The principal measurement from the study is clenching force as measured by the sensor relative to a maximum clenching force that is established via a calibration procedure for each user (i.e. force is report as a percentage value of maximum clenching force). The clenching force is sampled 4 times per second while worn by a user resulting in a time series of data for each night of data for each user.
  From this data two additional measurements are derived to establish the frequency of bruxing events. The first a measure of clenching events, defined as a measurement exceeded 10% of maximum bruxing force during at least one sample. The second measurement is total clenching time, which is defined as the aggregate time where the user exceeds a clenching force of 10% for one night of data.

CONTACTS AND LOCATIONS:
Locations (1):
- Otis Dental, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No